CLINICAL TRIAL: NCT05797974
Title: Does a Virtual Coach Offer a Better Solution for Weight Reduction in Ventral Hernia Patients With Obesity?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202300391; UL1TR001427 (NIH)
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Ventral Hernia
MeSH Terms: conditions — Obesity; Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual coach (Experimental): Participants will utilize the MyChart enabled virtual coach to aid preoperative weight loss.
  Interventions: Other: MyChart enabled virtual weight loss coach
- Standard weight loss tools (Active Comparator): Participants will not utilize the MyChart enabled virtual coach to aid preoperative weight loss, but instead use standard weight loss tools.
  Interventions: Other: Standard preoperative weight loss tools

INTERVENTIONS:
Other: MyChart enabled virtual weight loss coach — MyChart-enabled virtual coach utilized to aid in preoperative weight loss.
  Arms: Virtual coach
Other: Standard preoperative weight loss tools — Participants will utilize current standard preoperative weight loss tools.
  Arms: Standard weight loss tools

SUMMARY:
The purpose for this research is to create a MyChart-enabled virtual coach that assists obese patients lose weight prior to ventral hernia surgery. Researchers intend to show how the use of a virtual coach is more effective in preoperative weight reduction prior to ventral hernia repair over usual care. Correspondingly, this may lower unplanned hospital readmissions. For this clinical trial, where randomization is not possible, the study team will implement the use of propensity score matching that sorts individuals into different study arms as if randomly assigned. The primary outcome is the average net amount of time-dependent weight change per group over six months. Secondary outcomes are for the intervention group, patient satisfaction with the virtual coach and for both groups, quality of life. In addition, areas of social and economic disadvantage will be identified that may contribute to higher obesity rates. Machine learning (ML) modeling will be used to determine the important features for weight lost over the course of the study. The impact of this work will be to demonstrate efficacy and realized workflow efficiencies within a hospital-based surgery clinic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 90 years of age with a Body Mass Index (BMI) of 30 and above and diagnosed with Obesity by the ICD 10 Code: E66.9 who have been evaluated by a surgeon and offered elective ventral hernia repair. Also, participants must have a complete medical record that allows for all statistical calculations to be performed.

Exclusion Criteria:

* Pregnant females, patients with severe mental disorders, prescribed psychiatric medications associated with weight gain, a history of a Substance Use Disorder, patients on long-term steroid therapy, and patients with insufficient medical records.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jana Sacco, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled February 15, 2024 in ambulatory surgical clinic.
Pre-assignment Details: Of 33 enrolled participants, 32 met inclusion criteria and were included in study participation.
Period: Overall Study
Arm/Group | Virtual Coach | Standard Weight Loss Tools
Started | 28 | 4
Completed | 3 | 1
Not Completed | 25 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Coach | Standard Weight Loss Tools | Total
Number analyzed (Participants) | 28 | 4 | 32
Age, Continuous [Mean (Full Range); unit: years] | 50 [30 to 70] | 58 [30 to 70] | 51 [30 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 1 | 23
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 1 | 15
  White | 13 | 3 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 45 [34 to 60] | 40 [34 to 60] | 44 [34 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Pounds of Weight Change Per Group
Description: Average net amount of weight change
Time Frame: 6 months
Population: Intent to treat population (all participants assigned to virtual coach or standard weight loss tool)
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Virtual Coach | Standard Weight Loss Tools
Number analyzed (Participants) | 28 | 4
lbs | 24.25 (9.95) | 24.25 (9.95)

2. Secondary Outcome: Number of Interactions
Description: number of interactions with virtual coach per subject; interactions were determined as a digital responses logged from participants in the electronic medical record (MyChart)
Time Frame: 6 months
Population: 3 of the 25 virtual coach participants completed the 6 month survey
Measure: Mean (Full Range); unit: number of interactions
Arm/Group | Virtual Coach
Number analyzed (Participants) | 3
number of interactions | 9 [0 to 10]

3. Secondary Outcome: Degree of Quality of Life
Description: quality of life measured per the Hernia Related Quality of Life Survey (HerQLes), a validated self-reported 12-question tool used to assess the impact of a ventral hernia on a patient's quality of life and abdominal wall function. The tool helps measure a patient's quality of life before and after a ventral hernia repair (VHR). Scores are converted to a 0-100 scale, with higher scores indicating a better quality of life.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Coach | Standard Weight Loss Tools
Number analyzed (Participants) | 28 | 4
score on a scale | 46.19 (18.11) | 46.19 (18.11)

4. Secondary Outcome: Degree of Satisfaction With the Virtual Coach
Description: Satisfaction with the virtual coach will be measured by a single question, "How satisfied are you with the virtual coach." and rated on a 7 point Likert scale, from 1, Not satisfied at all, 4 Neutral to 7, Very satisfied.
Time Frame: 6 months
Population: Insufficient participation in 6 month survey to calculate degree of significance for outcome measure.
Measure: Number; unit: score on a scale
Arm/Group | Virtual Coach
Number analyzed (Participants) | 1
score on a scale | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Virtual Coach | Standard Weight Loss Tools
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/4
Other Adverse Events (participants affected / at risk) | 0/28 | 0/4

LIMITATIONS AND CAVEATS:
Insufficient participation in 6 month surveys to calculate degree of significance for outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT05797974/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT05797974/ICF_000.pdf